CLINICAL TRIAL: NCT00001089
Title: Human Immunodeficiency Virus (HIV) and Cytomegalovirus (CMV) Viral Burden and Development of CMV End-Organ Disease: A Prospective Study in HIV-Infected Individuals.
Brief Title: A Study of HIV and Cytomegalovirus (CMV) in HIV-Infected Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 360
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-02

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Prospective Studies; HIV-1; Cytomegalovirus; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Anti-HIV Agents; Viral Load; Multiple Organ Failure
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Acquired Immunodeficiency Syndrome; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To define relationships between 1) HIV load and risk of CMV disease, 2) CMV load and the risk of developing CMV disease, and 3) CMV load and HIV load. To establish threshold CMV and HIV load values in peripheral blood fractions that are associated with development of CMV end-organ disease. To define the natural history of CMV diseases in the context of highly active antiretroviral therapy (HAART).

Establishment of threshold CMV and HIV load values associated with CMV disease would facilitate identification of HIV-infected individuals truly at risk for CMV disease in whom targeted prophylactic interventions to prevent CMV disease would be indicated. These studies would also further the understanding of the natural history of CMV disease within the context of AIDS. Natural history studies conducted prior to the advent of highly active antiretroviral therapy (HAART; i.e., 3-drug regimens that include HIV reverse transcriptase and protease inhibitors) have demonstrated that the risk for developing CMV disease increases with progression of HIV disease and with declining CD4 counts. Presently the need exists to define the natural history of CMV disease in patients with AIDS within the context of HAART.

DETAILED DESCRIPTION:
Establishment of threshold CMV and HIV load values associated with CMV disease would facilitate identification of HIV-infected individuals truly at risk for CMV disease in whom targeted prophylactic interventions to prevent CMV disease would be indicated. These studies would also further the understanding of the natural history of CMV disease within the context of AIDS. Natural history studies conducted prior to the advent of highly active antiretroviral therapy (HAART; i.e., 3-drug regimens that include HIV reverse transcriptase and protease inhibitors) have demonstrated that the risk for developing CMV disease increases with progression of HIV disease and with declining CD4 counts. Presently the need exists to define the natural history of CMV disease in patients with AIDS within the context of HAART.

In this prospective observational study, HIV-infected patients who are CMV-seropositive with no clinical symptoms of CMV disease at entry are followed for three years or until the diagnosis of CMV end-organ disease or death, whichever comes first. Clinical evaluations are performed at baseline and every 8 weeks. Blood samples for virologic studies are taken every 16 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antivirals with anti-CMV activity (such as acyclovir, ganciclovir, valacyclovir, valganciclovir, foscarnet, etc.) for reasons other than treatment of CMV disease.
* Antivirals for prophylaxis or treatment of other herpesvirus infections.

Patients must have:

* Documented HIV-1 infection.
* Documented evidence of CD4 count <= 50 cells/mm3 in the previous 24 months.
* Presence of serum CMV IgG antibodies.
* No history of CMV end-organ disease or evidence of active CMV disease prior to study entry. NOTE: A history of positive CMV urine or blood cultures is acceptable as long as it has been determined that the patient does not have CMV end-organ disease.
* Signed, informed consent of parent or legal guardian for patients less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Ocular media opacities that preclude adequate visualization of the fundi.

Patients with the following prior conditions are excluded:

* History of CMV end-organ disease.
* Any pre-existing necrotizing retinopathy that may interfere with a subsequent diagnosis of CMV retinitis.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400

CONTACTS AND LOCATIONS:
Overall Officials: Erice A, Study Chair; Hirsch M, Study Chair; Polsky B, Study Chair
Locations (36):
- United States (36):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Children's Hosp of Denver, Denver, Colorado
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - St Vincent's Hosp / Mem Sloan-Kettering Cancer Ctr, New York, New York
  - Community Health Network Inc, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee